CLINICAL TRIAL: NCT05317026
Title: Pre-irradiation Vertebroplasty in Patients With Spine Metastases Candidates for SBRT vs SBRT Alone: Increased Early Pain Relief
Brief Title: Increased Early Pain Relief by Adding Vertebroplasty to SBRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-10542
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Spine Metastases; Radiation Therapy; Pain
MeSH Terms: conditions — Pain | interventions — Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-SBRT (Experimental): Vertebroplasty followed by Stereotactic Body Radiation Therapy (SBRT)
  Interventions: Procedure: Vertebroplasty
- SBRT (Other): SBRT is the actual standard of care.
  Interventions: Procedure: Stereotactic Body Radiation Therapy only

INTERVENTIONS:
Procedure: Vertebroplasty — SBRT consists of radiotherapy treatments hypofractionated in 1 to 5 fractions, at doses considered curative at a precise target volume.
  The vertebroplasty will be performed according to the usual procedure at the center in the angiography suite under local anesthesia and conscious sedation
  * Introduction of a vertebral needle, under biplanar fluoroscopic guidance, polymethylmethacrylate (PMMA) cement injection.
  * Cone-beam volume-CT at the end of the procedure, with the angiography table and c-arm, to evaluate the cement distribution and detect any leak.
  * Decubitus position for 2 hours following procedure, then hospital discharge on the same day.
  Arms: V-SBRT
Procedure: Stereotactic Body Radiation Therapy only — SBRT consists of radiotherapy treatments hypofractionated in 1 to 5 fractions, at doses considered curative at a precise target volume
  Other Names: SBRT
  Arms: SBRT

SUMMARY:
The goal of treating metastases is to preserve stability and neurological function while reducing pain. The actual standard of care is stereotaxic body radiation therapy (SBRT) alone in non-surgical patients. The added value of vertebroplasty to SBRT is not well documented in the literature, nor whether performing vertebroplasty before radiotherapy treatment leads to a reduction in the rate of fractures and post-SBRT pain.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of cancer.
* Spinal and vertebral bone metastases (T5 to L5) documented by imaging.
* Pain related to metastases ≥ 4 on a numerical scale 0-10.
* Karnofsky performance index > 60 (ecog 0-2)
* Candidate for SBRT
* Less than 3 consecutive levels reached.
* Ability to complete follow-up questionnaires regarding pain, analgesics, and quality of life assessment.
* Potentially unstable lesions according to the spinal instability neoplastic score (SINS) scale (> or = 7)

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Contraindications to MRI.
* Histology: myeloma, lymphoma or plasmacytoma.
* Radiotherapy prior to the level to be treated.
* Previous surgery at the site to be treated.
* Surgical indication:

spinal instability neoplastic score (SINS) > 13 or according to tumor board consensus.

Bilsky score > or = 2 Severe or progressive neurological signs (motor, incontinence).

* Lesion too large for safe vertebroplasty.
* High thoracic location not allowing safe visibility in fluoroscopy to perform vertebroplasty (T4 and above).
* Non-reversible coagulation disorders.
* Uncontrolled local or systemic infection.
* Estimated survival of less than 6 months.
* Inability or refusal to undergo SBRT treatment or vertebroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain change at 1 month | 1 month following the treatment
  Visual Analogue Scale, from 0 to 10, 10 being the highest pain

SECONDARY OUTCOMES:
Pain change | 1 week, 1 month, 3 months and 6 months post treatment
  Visual Analogue Scale, from 0 to 10, 10 being the highest pain
Change in level of physical, psychological and social functions | at 1 week, 1 month, 3 months and 6 months post treatment
  EORTC Quality of life Questionnaire : QLQ-C30 (score between 0 and 100, highest numbers represents higher response and quality of life)
Change in symptoms related to bone metastasis | at 1 week, 1 month, 3 months and 6 months post treatment
  QLQ-Bone metastases : BM22 questionnaire (All of the scales range in score from 0 to 100. A high score for the symptom scales represents a high level of symptomatology or problems, whilst a high score for the functional scales represents a high level of functioning)
Change in performance for activities of daily living | at 1 week, 1 month, 3 months and 6 months post treatment
  Karnofsky performance scale (score from 0 to 100, the lower the Karnofsky score, themore disable the patient is and need assistance)
Post-treatment fracture rates | at 3, 6, 12 and 24 months post treatment
  evaluation by MRI +/- CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Freire, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - Véronique Freire, Montreal, Quebec